CLINICAL TRIAL: NCT06845371
Title: MELODY Registry Follow-Up Study
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Melody
Record Dates: First submitted 2025-02-07; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease (CHD)
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Extension of the MELODY Registry, to assess longterm follow-up clinical results of Melody valve implantation after its commercialization in Europe / OUS

ELIGIBILITY:
Inclusion Criteria:

* previous inclusion in the MELODY Registry

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent Melody valve implantation into the pulmonary position after its commercialization in Europe / OUS
Sampling Method: Probability Sample
Enrollment: 845 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
primary outcome | from december 2006 up to December 2027
  • composite endpoint of TPVI related follow-up events (i.e. death, reoperation, or reintervention >48h after TPVI)

SECONDARY OUTCOMES:
secondary measure | from december 2006 up to December 2027
  TPVI infective endocarditis (I.E.) according to modified Duke criteria n

IPD SHARING:
Plan to Share IPD: Undecided